CLINICAL TRIAL: NCT03758781
Title: The IRX-2 Regimen Combined With Nivolumab in Recurrent/Metastatic Solid Tumors: A Phase 1b Study to Evaluate the Safety, Determine Recommended Phase 2 Dose (RP2D), and Investigate the Biologic and Clinical Activity
Brief Title: IRX-2 Regimen Combined With Nivolumab in Recurrent/Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19491
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Cancer; Recurrent Cancer; Solid Tumor; Renal Cell Carcinoma; Urothelial Carcinoma; NSCLC; Squamous Cell Carcinoma; Non-Small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Carcinoma, Squamous Cell; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — IRX 2; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IRX-2 Regimen combined with Nivolumab (Experimental): IRX-2 Regimen (4 ml) combined with Nivolumab (240 mg)
  Interventions: Drug: IRX 2; Drug: Nivolumab

INTERVENTIONS:
Drug: IRX 2 — IRX-2 Regimen: 21 day regimen of cyclophosphamide on Day 1 and subcutaneous IRX-2 injections for 10 days between Days 4 and 18. This 21 day regimen will be given every 12 weeks.
Drug: Nivolumab — Nivolumab 240 mg will be given via IV infusion once every 2 weeks.

SUMMARY:
This study is to determine the safety of IRX-2 Regimen combined with Nivolumab in patients with recurrent metastatic solid tumors. Researchers believe that this combination will have a tolerable safety profile and will increase the response rate in comparison to Nivolumab alone.

DETAILED DESCRIPTION:
The first phase of this trial is to establish the safety of IRX-2 Regimen combined with Nivolumab. The IRX-2 Regimen is a 21-day regimen of cyclophosophamide on Day 1 and subcutaneous IRX-2 injections for 10 days between Days 4 and 18. If no dose limiting toxicities (DLTs) are observed during the first 4 weeks of treatment, the enrollment will continue in a dose expansion phase. If there is a study treatment related DLT in 1 of 6 patients, the same dose will be investigated at the dose expansion cohorts. If study treatment related DLT is observed in 2 of 6 patients, accrual will be stopped and new dose levels or treatment sequences will be considered.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Participants must have histologically or cytologically confirmed renal cell carcinoma,urothelial carcinoma, non-small cell lung cancer, squamous cell carcinoma of the head and neck or melanoma.
* Participants must have recurrent or metastatic disease that is not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
* Must be willing and able to give informed consent and adhere to protocol therapy; written informed consent and any locally required authorization must be obtained from the participant prior to performing any protocol-related procedures, including screening evaluations
* Prior exposure to PD-1/PD-L1 inhibitor monotherapy, or prior exposure to CTLA-4 inhibitor monotherapy is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate normal organ and marrow function
* Participants who are receiving therapeutic anti-coagulant therapy are eligible.
* Palliative radiation therapy is allowed to non-target lesions at the discretion of the treating physician.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1.
* Life expectancy of greater than 3 months.
* Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to treatment.
* Body weight must be greater than 66 pounds.

Exclusion Criteria:

* Prior exposure to a combination of IRX-2 regimen, PD-1/PD-L1 inhibitors and CTLA-4 inhibitors are excluded. Prior exposure to PD-1/PD-L1 inhibitors is allowed.
* Radiation therapy with a curable intent within 30 days of first dose of study treatment is excluded. However, radiation therapy with a palliative intent is allowed to treat after 14 days from the last dose of radiation.
* Any medical contraindications or previous therapy that would preclude treatment with the IRX-2 Regimen, or nivolumab.
* Any unresolved toxicity Grade 2 or greater from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with IRX-2, or nivolumab may be included only after consultation with the study physician.
* Active or prior documented autoimmune or inflammatory disorders
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study treatment. Some exceptions apply.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Symptomatic cardiopulmonary disease, coronary artery disease, serious arrhythmia or chronic lung disease. Participants with these conditions who are stable with relatively minor symptoms and who are appropriate candidates for systemic treatments need not be excluded.
* Myocardial infarction within the last 3 months.
* Known infection with hepatitis B, hepatitis C, or HIV.
* Signs or symptoms of systemic infection (use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection).
* Clinically significant gastritis or peptic ulcer disease
* Stroke or other symptoms of cerebral vascular insufficiency within the last 3 months.
* Allergy to ciprofloxacin (or other quinolones).
* Previous diagnosis of invasive cancer from which the individual is not disease-free AND that has required treatment within the past 3 years, except for superficial skin, cervical cancer in-situ, or early stage prostate or bladder cancer (i.e. treatment with curative intent and long term disease-free expectations).
* History of leptomeningeal carcinomatosis
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ effective birth control from screening to 1 year after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience Dose Limiting Toxicities (DLTs) | Up to Day 28
  A DLT is defined as any Grade 3 or higher toxicity which occurs during the DLT evaluation period of 4 weeks (during Cycle 1 Day 1 and Cycle 1 Day 28) and considered related to study treatment. Toxicity that is clearly and directly related to the primary disease or to another etiology is excluded.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 12 months
  Objective response determined using Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 and Immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria.
Progression Free Survival of combination therapy | Up to 12 months
  Progression free survival defined as the time from Day 1 of treatment to evidence of progression. Progression will be defined by RECIST Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Jain, MD, MPH, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States